CLINICAL TRIAL: NCT03035214
Title: Single Arm Study on Treatment Algorithm to Justify Steroid Use in Selected Preterm Neonates to Prevent Bronchopulmonary Dysplasia
Brief Title: Study to Justify Steroid Use in Preterm Neonates to Prevent Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maadi Military Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Wael Hamza, Principal investigator, Maadi Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MaadiPed001
Record Dates: First submitted 2017-01-22; First posted 2017-01-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Dexamethasone; Steroids

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention of dysplasia through steroids (Other): Failure of lung tolerance to oxygen reduction will be defined as oxygen saturation 80 to 87% for 5 minutes, or <80% for 1 minute, then inspired oxygen will be increased back to the base line. This will be considered as an early predictor of evolving bronchopulmonary dysplasia. If there is no hypoventilation, dexamethasone will be given 0.25 mg/ kg/ d divided twice for 5 days intravenous.
  Interventions: Drug: Dexamethasone (Steroids)

INTERVENTIONS:
Drug: Dexamethasone (Steroids) — Is to describe the use of integrated assessment of respiratory physiology using Targeted Neonatal Echocardiography, assessment of optimal Functional Residual Capacity and the tolerance of lung oxygen uptake at different oxygen levels, and hence early prediction of Bronchopulmonary Dysplasia and the underlying pathophysiology by periodic application of the oxygen tolerance test; which may help early targeted treatment of this common disease.
  Other Names: Dexamethasone

SUMMARY:
Most preterm babies require supplemental oxygen for a variable period of time, up to several weeks or months after birth. The aim of oxygen therapy is to achieve adequate oxygen supply to the tissues without causing oxygen toxicity and oxidative stress. The current routine monitoring relies on oxygen saturation by pulse oximetry without identifying the underlying pathology, as lung parenchyma and pulmonary vascular disease can be contributed in pathophysiology at variable degrees.

Steroids usage for prevention of Bronchopulmonary dysplasia also has been shown to have adverse neurodevelopmental outcome. Available data are conflicting and inconclusive; clinicians must use their own clinical judgment to balance the adverse effects of Bronchopulmonary dysplasia with the potential adverse effects of treatments for each individual patient. Very low birth weight infants who remain on mechanical ventilation after 1 to 2 weeks of age are at very high risk of developing Bronchopulmonary dysplasia.

When considering corticosteroid therapy for such an infant, clinicians might conclude that the risks of a short course of glucocorticoid therapy to prevent Bronchopulmonary dysplasia are warranted.

DETAILED DESCRIPTION:
This is a prospective study. 30 Preterm infants admitted to neonatal intensive care units of Maadi, Ghamra military hospitals, and Ain Shams University hospitals, will be prospectively enrolled within 24 hours after birth. Daily evaluation of oxygen histograms with measurement of the cumulative time of oxygen saturations below 80%, (risk of hypoxemia and potential tissue hypoxia), and arterial oxygen saturations Sao2 above 95% (potential risk of hyperoxia and increased oxidative stress). Evaluation window will be on a weekly basis as long as the infant is on oxygen support and by applying oxygen tolerance test. The treating clinical team will be blinded to all results of Oxygen tolerance test.

ELIGIBILITY:
All preterm neonates admitted to the neonatal intensive care unit will be considered eligible for inclusion. Fully informed written consent from parents of all eligible infants will be sought prior to enrollment. Infants with major congenital abnormalities, cardiac lesions other than Patent ductus arteriosus, and lung hypoplasia will be excluded from this study.

Inclusion criteria:

* < 36 week gestation pre-terms, not having major congenital anomalies

Exclusion criteria:

* Congenital heart disease
* Major congenital abnormalities

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-02-19 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant morbidity | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Maadi Military Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No